CLINICAL TRIAL: NCT04697316
Title: Transcranial Direct Current Stimulation (tDCS) as a Cognitive Functioning Enhancement Treatment for ADHD Patients Compared to Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Noa Beiman, Principal Investigator, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tDCS-ADHD
Record Dates: First submitted 2020-12-31; First posted 2021-01-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Transcranial Direct Current Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADHD tDCS (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation
- ADHD Sham (Sham Comparator)
  Interventions: Device: Sham
- Healthy control tDCS (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation
- Healthy control Sham (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — To stimulate the left DLPFC, the anode electrode will be placed over F3 and the cathode will be placed over F4. Each stimulation will be applied for 20 min at 2mA intensity.
  Arms: ADHD tDCS; Healthy control tDCS
Device: Sham — For the sham treatment, stimulation will be stopped after 30 seconds. Current will be renewed five times throughout the session for 2 seconds each time, to mimic the tDCS stimulation.
  Arms: ADHD Sham; Healthy control Sham

SUMMARY:
This study will examine the possible effects of tDCS (Transcranial Direct Current Stimulation) treatment to the left DLPFC on cognitive functions which were found to be deficient amongst ADHD patients. The study will include 100 subjects, 50 of whom diagnosed with ADHD. Subjects will complete the ASRS questionnaire to measure ADHD symptoms severity. Next, subjects will complete a series of cognitive tasks, after which they will receive either tDCS treatment or a sham treatment. Finally, subjects will repeat the cognitive tasks. Later that day, a telephonic follow up will take place. ADHD symptoms will be assessed again the next day.

ELIGIBILITY:
Inclusion Criteria:Participation criteria for healthy participants

1. Right hand dominance.
2. No psychiatric nor neural diagnosis.
3. Participants must be able to comprehend the study's procedure and sign an informed consent.

Participation criteria for ADHD diagnosed participants

1. ADHD diagnosis (according to DSM V).
2. Right hand dominance.
3. Participants must be able to comprehend the study's procedure and sign an informed consent.
4. Participants who regularly use Methylphenidate will be required to avoid the medication for 24 hours prior to study and 12 hours post study.

   -

Exclusion Criteria:

* a. Other psychiatric diagnoses (additional to ADHD). b. Drug use (excluding Methylphenidate). c. Neurological disorders. d. Pacemaker, Insulin pump

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
N-back | through study completion
  change in working memory: increase in hit rate
Stroop | through study completion, up to 1 hour after treatment
  change in interference control: smaller interference effect
Stop-signal | through study completion, up to 1 hour after treatment
  change in response inhibition: shorter SSRT
Time Reproduction task | through study completion, up to 1 hour after treatment
  change in time perception: increased accuracy
Continuous Performance Task | through study completion, up to 1 hour after treatment
  change in continuous concentration: increase in accuracy
Navon task | through study completion, up to 1 hour after treatment
  change in accuracy, shorter RT's

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No